CLINICAL TRIAL: NCT02746445
Title: A Longitudinal Study on the Safety and Efficacy for Subjects With Autism Spectrum Disorder (ASD) Who Received Magnetic EEG/ECG-Guided Resonance Therapy (MeRT)
Brief Title: A Longitudinal Study on the Safety and Efficacy for Subjects With ASD Who Received MeRT
Status: Completed | Type: Observational
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Other Study IDs: MeRT-015
Record Dates: First submitted 2016-04-15; First posted 2016-04-21 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Autistic Disorder
Keywords: Autism; ASD; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ASD Subjects: No interventions. This is an observation of subjects who received MeRT utilizing assessment documentation.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. This is a longitudinal study looking at subjects who received MeRT treatment.
  Other Names: No intervention.

SUMMARY:
The purpose of this study is to continue to evaluate the long-term effectiveness of Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) in children with Autism Spectrum Disorder (ASD). No active MeRT treatment will be performed in this study.

DETAILED DESCRIPTION:
This clinical trial is a longitudinal study designed to evaluate the safety and efficacy for subjects with Autism Spectrum Disorder (ASD) who received Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) in the IRB approved clinical trial. A total of twenty-eight (28) subjects will be followed in this study. After providing informed consent, twenty-eight (28) subjects who participated in the previous protocol will be observed for up to three (3) years post-MeRT treatment. During this period, subjects will be evaluated at 104 and 156 weeks post-MeRT treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have completed the MeRT-001 (formerly known as MRT-001) clinical trial conducted by the Brain Treatment Center (BTC)
2. Age between 6 and 15 years (at day of informed consent)
3. Willing and able to adhere to the study visits

Exclusion Criteria:

1. Subjects who did not participate in the MeRT-001 clinical trial.
2. Any condition which in the judgment of the investigator would prevent the subject from completion of the study.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Twenty-eight (28) male and female individuals diagnosed with Autism Spectrum Disorder (ASD) who participated in the initial treatment protocol will be followed.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in Childhood Autism Rating Scale (CARS) | Change from baseline CARS score at 104 weeks post-MeRT treatment
  Symptom reduction in ASD will be measured using the arithmetic reduction in the CARS total score between two time points BL and week 104 (or Early Termination)

SECONDARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | Baseline, weeks 5, 10, and 12, and 104 and 156 weeks post-MeRT treatment
  Symptom reduction in ASD will be measured using the arithmetic reduction in the CARS total score between the multiple time points of the MeRT-001 trial (BL, Week 5, 10 and 12), BL, Follow-Up 1 Post-MeRT Treatment (Week 104), and Follow-Up 2 Post-MeRT Treatment (Week 156).

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Young Kim, MD, Principal Investigator — Brain Treatment Center
Locations (1):
- Brain Treatment Center, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Betancur C, Sakurai T, Buxbaum JD. The emerging role of synaptic cell-adhesion pathways in the pathogenesis of autism spectrum disorders. Trends Neurosci. 2009 Jul;32(7):402-12. doi: 10.1016/j.tins.2009.04.003. Epub 2009 Jun 21. PMID 19541375
- [Background] Crespi B, Stead P, Elliot M. Evolution in health and medicine Sackler colloquium: Comparative genomics of autism and schizophrenia. Proc Natl Acad Sci U S A. 2010 Jan 26;107 Suppl 1(Suppl 1):1736-41. doi: 10.1073/pnas.0906080106. Epub 2009 Dec 1. PMID 19955444
- [Background] Stigler KA, S.T., Posey DJ, McDougle CJ, Autism and immune factors: a comprehensive review. Res Autism Spectr Disord 3(4): 840-860. 2009.
- [Background] Krakowiak P, Walker CK, Bremer AA, Baker AS, Ozonoff S, Hansen RL, Hertz-Picciotto I. Maternal metabolic conditions and risk for autism and other neurodevelopmental disorders. Pediatrics. 2012 May;129(5):e1121-8. doi: 10.1542/peds.2011-2583. Epub 2012 Apr 9. PMID 22492772
- [Background] Levy SE, Mandell DS, Schultz RT. Autism. Lancet. 2009 Nov 7;374(9701):1627-38. doi: 10.1016/S0140-6736(09)61376-3. Epub 2009 Oct 12. PMID 19819542
- [Background] Just MA, Cherkassky VL, Keller TA, Kana RK, Minshew NJ. Functional and anatomical cortical underconnectivity in autism: evidence from an FMRI study of an executive function task and corpus callosum morphometry. Cereb Cortex. 2007 Apr;17(4):951-61. doi: 10.1093/cercor/bhl006. Epub 2006 Jun 13. PMID 16772313
- [Background] Buie T, Campbell DB, Fuchs GJ 3rd, Furuta GT, Levy J, Vandewater J, Whitaker AH, Atkins D, Bauman ML, Beaudet AL, Carr EG, Gershon MD, Hyman SL, Jirapinyo P, Jyonouchi H, Kooros K, Kushak R, Levitt P, Levy SE, Lewis JD, Murray KF, Natowicz MR, Sabra A, Wershil BK, Weston SC, Zeltzer L, Winter H. Evaluation, diagnosis, and treatment of gastrointestinal disorders in individuals with ASDs: a consensus report. Pediatrics. 2010 Jan;125 Suppl 1:S1-18. doi: 10.1542/peds.2009-1878C. PMID 20048083
- [Background] Happe F, Ronald A. The 'fractionable autism triad': a review of evidence from behavioural, genetic, cognitive and neural research. Neuropsychol Rev. 2008 Dec;18(4):287-304. doi: 10.1007/s11065-008-9076-8. Epub 2008 Oct 28. PMID 18956240
- [Background] Amaral DG, Schumann CM, Nordahl CW. Neuroanatomy of autism. Trends Neurosci. 2008 Mar;31(3):137-45. doi: 10.1016/j.tins.2007.12.005. Epub 2008 Feb 6. PMID 18258309
- [Background] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818
- [Background] Billstedt E, Gillberg IC, Gillberg C. Autism after adolescence: population-based 13- to 22-year follow-up study of 120 individuals with autism diagnosed in childhood. J Autism Dev Disord. 2005 Jun;35(3):351-60. doi: 10.1007/s10803-005-3302-5. PMID 16119476
- [Background] Langstrom N, Grann M, Ruchkin V, Sjostedt G, Fazel S. Risk factors for violent offending in autism spectrum disorder: a national study of hospitalized individuals. J Interpers Violence. 2009 Aug;24(8):1358-70. doi: 10.1177/0886260508322195. Epub 2008 Aug 13. PMID 18701743
- [Background] Posey DJ, Stigler KA, Erickson CA, McDougle CJ. Antipsychotics in the treatment of autism. J Clin Invest. 2008 Jan;118(1):6-14. doi: 10.1172/JCI32483. PMID 18172517
- [Background] Happe F, Ronald A, Plomin R. Time to give up on a single explanation for autism. Nat Neurosci. 2006 Oct;9(10):1218-20. doi: 10.1038/nn1770. PMID 17001340
- [Background] Larsson HJ, Eaton WW, Madsen KM, Vestergaard M, Olesen AV, Agerbo E, Schendel D, Thorsen P, Mortensen PB. Risk factors for autism: perinatal factors, parental psychiatric history, and socioeconomic status. Am J Epidemiol. 2005 May 15;161(10):916-25; discussion 926-8. doi: 10.1093/aje/kwi123. PMID 15870155
- [Background] Geschwind DH. Autism: many genes, common pathways? Cell. 2008 Oct 31;135(3):391-5. doi: 10.1016/j.cell.2008.10.016. PMID 18984147
- [Background] Hultman CM, Sparen P, Cnattingius S. Perinatal risk factors for infantile autism. Epidemiology. 2002 Jul;13(4):417-23. doi: 10.1097/00001648-200207000-00009. PMID 12094096
- [Background] Cheslack-Postava K, Liu K, Bearman PS. Closely spaced pregnancies are associated with increased odds of autism in California sibling births. Pediatrics. 2011 Feb;127(2):246-53. doi: 10.1542/peds.2010-2371. Epub 2011 Jan 10. PMID 21220394
- [Background] Sebat J, Lakshmi B, Malhotra D, Troge J, Lese-Martin C, Walsh T, Yamrom B, Yoon S, Krasnitz A, Kendall J, Leotta A, Pai D, Zhang R, Lee YH, Hicks J, Spence SJ, Lee AT, Puura K, Lehtimaki T, Ledbetter D, Gregersen PK, Bregman J, Sutcliffe JS, Jobanputra V, Chung W, Warburton D, King MC, Skuse D, Geschwind DH, Gilliam TC, Ye K, Wigler M. Strong association of de novo copy number mutations with autism. Science. 2007 Apr 20;316(5823):445-9. doi: 10.1126/science.1138659. Epub 2007 Mar 15. PMID 17363630
- [Background] Marshall CR, Noor A, Vincent JB, Lionel AC, Feuk L, Skaug J, Shago M, Moessner R, Pinto D, Ren Y, Thiruvahindrapduram B, Fiebig A, Schreiber S, Friedman J, Ketelaars CE, Vos YJ, Ficicioglu C, Kirkpatrick S, Nicolson R, Sloman L, Summers A, Gibbons CA, Teebi A, Chitayat D, Weksberg R, Thompson A, Vardy C, Crosbie V, Luscombe S, Baatjes R, Zwaigenbaum L, Roberts W, Fernandez B, Szatmari P, Scherer SW. Structural variation of chromosomes in autism spectrum disorder. Am J Hum Genet. 2008 Feb;82(2):477-88. doi: 10.1016/j.ajhg.2007.12.009. Epub 2008 Jan 17. PMID 18252227
- [Background] Weiss LA, Shen Y, Korn JM, Arking DE, Miller DT, Fossdal R, Saemundsen E, Stefansson H, Ferreira MA, Green T, Platt OS, Ruderfer DM, Walsh CA, Altshuler D, Chakravarti A, Tanzi RE, Stefansson K, Santangelo SL, Gusella JF, Sklar P, Wu BL, Daly MJ; Autism Consortium. Association between microdeletion and microduplication at 16p11.2 and autism. N Engl J Med. 2008 Feb 14;358(7):667-75. doi: 10.1056/NEJMoa075974. Epub 2008 Jan 9. PMID 18184952
- [Background] Ronald A, Happe F, Bolton P, Butcher LM, Price TS, Wheelwright S, Baron-Cohen S, Plomin R. Genetic heterogeneity between the three components of the autism spectrum: a twin study. J Am Acad Child Adolesc Psychiatry. 2006 Jun;45(6):691-699. doi: 10.1097/01.chi.0000215325.13058.9d. PMID 16721319
- [Background] Rogers SJ. What are infant siblings teaching us about autism in infancy? Autism Res. 2009 Jun;2(3):125-37. doi: 10.1002/aur.81. PMID 19582867
- [Background] Filipek PA, Accardo PJ, Baranek GT, Cook EH Jr, Dawson G, Gordon B, Gravel JS, Johnson CP, Kallen RJ, Levy SE, Minshew NJ, Ozonoff S, Prizant BM, Rapin I, Rogers SJ, Stone WL, Teplin S, Tuchman RF, Volkmar FR. The screening and diagnosis of autistic spectrum disorders. J Autism Dev Disord. 1999 Dec;29(6):439-84. doi: 10.1023/a:1021943802493. PMID 10638459
- [Background] Beaudet AL. Autism: highly heritable but not inherited. Nat Med. 2007 May;13(5):534-6. doi: 10.1038/nm0507-534. No abstract available. PMID 17479094
- [Background] Schmitz C, Rezaie P. The neuropathology of autism: where do we stand? Neuropathol Appl Neurobiol. 2008 Feb;34(1):4-11. doi: 10.1111/j.1365-2990.2007.00872.x. Epub 2007 Oct 26. PMID 17971078
- [Background] Piven J, Palmer P, Jacobi D, Childress D, Arndt S. Broader autism phenotype: evidence from a family history study of multiple-incidence autism families. Am J Psychiatry. 1997 Feb;154(2):185-90. doi: 10.1176/ajp.154.2.185. PMID 9016266
- [Background] Weissman JR, Kelley RI, Bauman ML, Cohen BH, Murray KF, Mitchell RL, Kern RL, Natowicz MR. Mitochondrial disease in autism spectrum disorder patients: a cohort analysis. PLoS One. 2008;3(11):e3815. doi: 10.1371/journal.pone.0003815. Epub 2008 Nov 26. PMID 19043581
- [Background] Frye RE, Melnyk S, Macfabe DF. Unique acyl-carnitine profiles are potential biomarkers for acquired mitochondrial disease in autism spectrum disorder. Transl Psychiatry. 2013 Jan 22;3(1):e220. doi: 10.1038/tp.2012.143. PMID 23340503
- [Background] Fournier KA, Hass CJ, Naik SK, Lodha N, Cauraugh JH. Motor coordination in autism spectrum disorders: a synthesis and meta-analysis. J Autism Dev Disord. 2010 Oct;40(10):1227-40. doi: 10.1007/s10803-010-0981-3. PMID 20195737
- [Background] Sigman M, Dijamco A, Gratier M, Rozga A. Early detection of core deficits in autism. Ment Retard Dev Disabil Res Rev. 2004;10(4):221-33. doi: 10.1002/mrdd.20046. PMID 15666338
- [Background] Sigman M, Spence SJ, Wang AT. Autism from developmental and neuropsychological perspectives. Annu Rev Clin Psychol. 2006;2:327-55. doi: 10.1146/annurev.clinpsy.2.022305.095210. PMID 17716073
- [Background] Iacoboni M, Dapretto M. The mirror neuron system and the consequences of its dysfunction. Nat Rev Neurosci. 2006 Dec;7(12):942-51. doi: 10.1038/nrn2024. Epub 2006 Nov 8. PMID 17115076
- [Background] Association, A.P., Diagnostic and statistical manual of mental disorders; DSM-IV. Vol. 4th. 2000.
- [Background] Johnson CP, Myers SM; American Academy of Pediatrics Council on Children With Disabilities. Identification and evaluation of children with autism spectrum disorders. Pediatrics. 2007 Nov;120(5):1183-215. doi: 10.1542/peds.2007-2361. Epub 2007 Oct 29. PMID 17967920
- [Background] Becker KG. Male gender bias in autism and pediatric autoimmunity. Autism Res. 2012 Apr;5(2):77-83. doi: 10.1002/aur.1227. Epub 2012 Mar 17. PMID 22431266
- [Background] Schopler E, Reichler RJ, DeVellis RF, Daly K. Toward objective classification of childhood autism: Childhood Autism Rating Scale (CARS). J Autism Dev Disord. 1980 Mar;10(1):91-103. doi: 10.1007/BF02408436. No abstract available. PMID 6927682
- [Background] Ozonoff S, Goodlin-Jones BL, Solomon M. Evidence-based assessment of autism spectrum disorders in children and adolescents. J Clin Child Adolesc Psychol. 2005 Sep;34(3):523-40. doi: 10.1207/s15374424jccp3403_8. PMID 16083393
- [Background] Schopler E, v.B.M., Wellman GJ, Love SR, CARS2 Childhood Autism Rating Scale, second edition. WPS Publishing: Torrance, CA. 2010.
- [Background] Helt M, Kelley E, Kinsbourne M, Pandey J, Boorstein H, Herbert M, Fein D. Can children with autism recover? If so, how? Neuropsychol Rev. 2008 Dec;18(4):339-66. doi: 10.1007/s11065-008-9075-9. Epub 2008 Nov 14. PMID 19009353
- [Background] Rogers SJ, Vismara LA. Evidence-based comprehensive treatments for early autism. J Clin Child Adolesc Psychol. 2008 Jan;37(1):8-38. doi: 10.1080/15374410701817808. PMID 18444052
- [Background] Seltzer MM, Shattuck P, Abbeduto L, Greenberg JS. Trajectory of development in adolescents and adults with autism. Ment Retard Dev Disabil Res Rev. 2004;10(4):234-47. doi: 10.1002/mrdd.20038. PMID 15666341
- [Background] Pickett E, Pullara O, O'Grady J, Gordon B. Speech acquisition in older nonverbal individuals with autism: a review of features, methods, and prognosis. Cogn Behav Neurol. 2009 Mar;22(1):1-21. doi: 10.1097/WNN.0b013e318190d185. PMID 19372766
- [Background] Magiati I, Charman T, Howlin P. A two-year prospective follow-up study of community-based early intensive behavioural intervention and specialist nursery provision for children with autism spectrum disorders. J Child Psychol Psychiatry. 2007 Aug;48(8):803-12. doi: 10.1111/j.1469-7610.2007.01756.x. PMID 17683452
- [Background] Fountain C, Winter AS, Bearman PS. Six developmental trajectories characterize children with autism. Pediatrics. 2012 May;129(5):e1112-20. doi: 10.1542/peds.2011-1601. Epub 2012 Apr 2. PMID 22473372
- [Background] MM, S., EEG Waves Classifier using wavelet Transform and Fourier Transform. International Journal of Medical, Pharmaceutical Science and Engineering, 1(3): p. 77 - 82. 2007.
- [Background] Roberts TP, Schmidt GL, Egeth M, Blaskey L, Rey MM, Edgar JC, Levy SE. Electrophysiological signatures: magnetoencephalographic studies of the neural correlates of language impairment in autism spectrum disorders. Int J Psychophysiol. 2008 May;68(2):149-60. doi: 10.1016/j.ijpsycho.2008.01.012. Epub 2008 Feb 12. PMID 18336941
- [Background] Kikuchi M, Yoshimura Y, Shitamichi K, Ueno S, Hirosawa T, Munesue T, Ono Y, Tsubokawa T, Haruta Y, Oi M, Niida Y, Remijn GB, Takahashi T, Suzuki M, Higashida H, Minabe Y. A custom magnetoencephalography device reveals brain connectivity and high reading/decoding ability in children with autism. Sci Rep. 2013;3:1139. doi: 10.1038/srep01139. Epub 2013 Jan 25. PMID 23355952